CLINICAL TRIAL: NCT05130034
Title: Home-based Pulmonary Rehabilitation and Health Coaching to Improve Respiratory-related Quality of Life and Physical Activity in Fibrotic Interstitial Lung Disease
Brief Title: Home-based Pulmonary Rehabilitation and Health Coaching in Fibrotic Interstitial Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Teng Moua, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-006804
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Fibrotic Interstitial Lung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based pulmonary rehab for fibrotic interstitial lung disease (Experimental): Subjects diagnosed with fibrotic interstitial lung disease will participate in a home-rehab program that promotes more physical activity in daily life.
  Interventions: Behavioral: Home-based pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Home-based pulmonary rehabilitation — Home-based tablet-assisted pulmonary rehabilitation with monitoring technology and telephonic health coach calls using motivational interviewing techniques

SUMMARY:
The purpose of this study is to gather information on the effectiveness of a home-based pulmonary rehabilitation program with health coaching and tele-monitoring for improving patient-reported respiratory-related quality of life and physical activity in patients with fibrotic Interstitial Lung Diseases (f-ILD).

DETAILED DESCRIPTION:
The home-based pulmonary rehabilitation program involves using a computer tablet paired with a pulse oximeter and activity tracker. Gentle upper body exercises, walking and a breathing practice are completed by following along on the computer tablet. Weekly check-in calls by telephone will be provided by a Health Coach to assess clinical status and monitor progress. The exercise portion of the program lasts 12 weeks. There are questionnaires and a research grade activity tracker measuring baseline and post-intervention findings at the end of 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis (IPF) or other fibrotic interstitial lung disease, with a minimum of > 10% fibrosis on computed tomography imaging.
* Clinically meaningful breathlessness: modified Medical Research Council (mMRC) dyspnea score >1.

Exclusion Criteria:

* Inability to walk (orthopedic/neurologic/cardiac limitation causing immobility).
* Cognitive impairment or inability to understand and follow instructions.
* Traditional PR completed within 3 months of study recruitment.
* Hospice or end-of-life care at the time of screening.
* Acute exacerbation at the time of screening.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported respiratory-related quality of life CRQ Physical Summary score | Baseline, 12 weeks
  Measured using the Chronic Respiratory Questionnaire (CRQ) survey which is a validated tool for measuring health status in patients with chronic lung disease divided into four domains of dyspnea, fatigue, emotion, and mastery. The Physical Summary score combines dyspnea and fatigue dimensions, a lower score suggests a greater degree of dysfunction on a 7-point scale. A difference of 0.5 in any domain is considered clinically significant (the minimal clinically important difference (MCID)). Higher total scores represent relatively better or improved patient-reported quality of life.
Change in patient-reported respiratory-related quality of life CRQ Emotional score | Baseline, 12 weeks
  Measured using the Chronic Respiratory Questionnaire (CRQ) survey which is a validated tool for measuring health status in patients with chronic lung disease divided into four domains of dyspnea, fatigue, emotion, and mastery. The emotional domain score is measured by a lower score suggests a greater degree of dysfunction on a 7-point scale. A difference of 0.5 in any domain is considered clinically significant (the minimal clinically important difference (MCID)). Higher total scores represent relatively better or improved patient-reported quality of life.
Physical activity | Baseline, 12 weeks
  Measured by mean number of steps per 24-hour period as assessed by Actigraphy, pre- and post-intervention

SECONDARY OUTCOMES:
Qualitative assessment of patient-reported efficacy | 12 weeks
  Measured at the end of study through qualitative interviews using structured interview guide, combined with primary outcomes using mixed-methods analysis. Potential themes of relevance being sought include changes in patient perception of disease severity, overcoming emotional and physical burden of disease, and feasibility and long-term utility of the intervention.
Self-reported tolerance of directed medical management | Baseline, 12 weeks
  Pre and post-intervention assessment of patient-reported side-effect severity from medical management

OTHER OUTCOMES:
Change in self-management ability | Baseline, 12 weeks
  Assessed pre and post-intervention using SMAS-30, a validated questionnaire highlighting six core self-management abilities including taking initiative, investment behavior, variety, multi-functionality, self-efficacy, and positive frame of mind. Higher total or domain scores suggest higher relative self-management ability.
Change in mood or affect | Baseline, 12 weeks
  Assessed pre and post-intervention using Positive and Negative Affect Scale (PANAS), a 20-item scale measures the positive and negative affective components of well-being. A ratio of 2.5 or higher for positive vs negative assessments suggests more positive mood.
Change in self-reported dyspnea | Baseline, 12 weeks
  Assessed pre and post-intervention using Modified Medical Research Council (mMRC) scale; a change in 1 point is the minimal clinically important difference (MCID), with HIGHER scores suggesting greater dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Teng Moua, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials